CLINICAL TRIAL: NCT06038669
Title: User Evaluation of a Home-collection Kit for People With Diabetes
Status: Recruiting | Type: Observational
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 3242
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with diabetes: Patients who have diabetes will be asked to use a home collection kit to collect a dried blood spot sample which will be compared to the HbA1C result.
  Interventions: Device: Dried blood spot device
- Health care professionals: Health care professionals who work with diabetic patients will be interviewed and asked about diabetes monitoring in the healthcare setting, comments on current laboratory service, patient engagement, comments on service improvement
  Interventions: Other: Healthcare professional interviews

INTERVENTIONS:
Device: Dried blood spot device — Patients will be asked to provide a dried blood spot sample
  Groups: People with diabetes
Other: Healthcare professional interviews — Health care professionals only will be interviewed using the topic guide and asked about their experience of diabetes monitoring
  Groups: Health care professionals

SUMMARY:
Type 1 and Type 2 are the most common types of diabetes mellitus. Although the cause of Type 1 is different to Type 2, they can both lead to high blood glucose levels as the patient is unable to store and use sugar. The disease is an epidemic of the 21st century which is increasing, having a current prevalence of approximately 8%.

Poor disease control is associated with a range of long-term health conditions which have a severe impact upon quality of life and are responsible for the increased morbidity and mortality associated with the disease.

Healthcare professionals use HbA1c as the main marker to monitor diabetic control. Patients with diabetes have regular review appointments to monitor their overall health and discuss their HbA1c target and results. The purpose of monitoring patients with diabetes is to improve patient outcomes. It is known that poor control is associated with poor clinical outcomes and also that reduced monitoring is linked to suboptimal diabetic control. Therefore, aiming for the correct monitoring frequency helps towards achieving the best control which can lead to the most favourable clinical outcomes. The inconvenience of attending for a blood test and follow-up appointment is a major factor affecting patient adherence to monitoring, locally approximately 50% of patients with diabetes have their HbA1c level measured either too soon or too late.

To address this issue and improve access to monitoring at the correct time interval we aim to produce a HbA1c home testing kit which can be posted back to the laboratory at the convenience of the patient. The kit will be developed based on feedback from patients with diabetes and will use a dried blood spot sample to produce HbA1c results comparable to the whole blood standard method.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type I or Type II diabetes
* Aged 18 years or over
* Venous blood sample for HbA1c collected within the two weeks prior to the clinic appointment
* Ability to provide fully informed consent

Exclusion Criteria:

* Non-English speaking where translation of the study documents and procedures could limit fully informed consent
* Severe visual impairment which would leave the participant unable to complete the study procedures.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetic patients (type I and II) aged over 18 years old.
  Healthcare professionals aged 18 or over who work with patients with diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
DBS kit assay performance | 1 year, 3 months
  For the DBS-based home collection kit used by patients to be 'fit for purpose', it must achieve the following:
  Assay performance - correlation and bias. Correlation coefficient (r2 value) from linear regression plot should be >0.95 with a bias of less than 5%.

SECONDARY OUTCOMES:
Participant questionnaires theme analysis | 1 year, 3 months
  Completed participant questionnaires will be collated and analysed for themes. We aim to determine whether participants deem the home-collection kit to be acceptable. The information gained will be used to design a full study.
Interviews | 1 year, 3 months
  The health care professional interview transcripts will be recorded and analysed. The emerging themes will be taken into consideration when designing the full study.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, United Kingdom

IPD SHARING:
Plan to Share IPD: No